CLINICAL TRIAL: NCT01948050
Title: Pilot Study on Safety and Efficacy of the Non-invasive Transcranial Stimulation (tDCS) to Relieve Neuropathic Pain in Cancer Patients
Brief Title: Pilot Study of Transcranial Stimulation (tDCS)to Relieve Neuropathic Pain in Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 038-08
Record Dates: First submitted 2013-08-20; First posted 2013-09-23 (Estimated); Results first posted 2014-07-14 (Estimated); Last update posted 2014-07-14 (Estimated); Status verified 2014-06

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- real tDCS stimulation (Experimental): non-invasive transcranial direct current stimulation (tDCS) at 2 milliamiampers (2mA)for 20 minutes at each session, on five consecutive days.
  Interventions: Device: non-invasive transcranial direct current stimulation (tDCS)
- Sham tDCS (Sham Comparator): sham non-invasive transcranial direct current stimulation (tDCS) consisting of 30 seconds of tDCS stimulation at 2mp and 19 minutes and 30 seconds of tdcs at 0mp stimulation,on five consecutive days.
  Interventions: Device: non-invasive transcranial direct current stimulation (tDCS)

INTERVENTIONS:
Device: non-invasive transcranial direct current stimulation (tDCS)

SUMMARY:
This is a pilot study designed to collect preliminary data on safety and efficacy of transcranial direct current stimulation (tDCS) to relieve pain in cancer patients who developed neuropathic pain in the affected area after a surgical intervention, radiation therapy, or chemotherapy to treat the disease.

DETAILED DESCRIPTION:
This is a pilot study that aims to determine the effect of repetitive tDCS stimulation, performed on five consecutive days at intensity of 2 mA, on pain and somatosensory abnormalities in patients with neuropathic pain that followed surgical, radiation or chemotherapeutic treatment, and to evaluate safety of tDCS in the same model.

ELIGIBILITY:
Adult male and female patients with cancer who developed neuropathic pain in the affected area secondary the surgical procedure, chemotherapy or radiation that meet the following Inclusion/Exclusion criteria:

Inclusion Criteria:

Pain on the side of the lesion

* Spontaneous pain with a score for "worst pain in the last 24 hours" >4 on a numeric scale 0-10
* Must present the following symptoms and signs:

  * Continuous burning, shooting, or lancinating pain.
  * Presence of hyperesthesia
  * Presence of hyperalgesia (to pinprick) and/or allodynia (to light touch)

Exclusion Criteria:

* Uncontrolled hypertension, uncontrolled diabetes, uncontrolled cardiovascular disease
* Pain/painful conditions unrelated to the cancer or related treatment
* Pregnancy
* History of seizures/epilepsy
* Any implanted devices (e.g. a cardio stimulator, etc)
* Active illegal drug/alcohol abuse
* Unable to follow directions or complete tools in English

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-01; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helena Knotkova, PhD, Principal Investigator — Beth Israel Medical Center
Locations (1):
- Beth Isael Medical Center, New York, USA, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 191 subjects identified. 33 were ineligible at pre-screening; 40 not reacahble; 21 lost to follow-up; 3 deceased; 56 not interested. 38 subjects consented.
Pre-assignment Details: 38 subjects consented; 8 screen failures; 6 never started; 24 were randomized. 1 subject withdrew after undergoing 4 of 5 tDCS/sham sessions. 23 completed randomized study.
Period: Overall Study
Arm/Group | Real tDCS Stimulation | Sham tDCS
Started | 16 | 8
Completed | 16 | 7
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Real tDCS Stimulation | Sham tDCS | Total
Number analyzed (Participants) | 16 | 8 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 8 | 21
  >=65 years | 3 | 0 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.9 (9.4) | 49.8 (13.4) | 54.5 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 11
  Male | 9 | 4 | 13
Region of Enrollment [Number; unit: participants]
  United States | 16 | 8 | 24

OUTCOME MEASURES:

1. Primary Outcome: Pain Intensity
Description: Measured on the 11 point numerical paid rating scale with anchor points 0 = no pain and 10 = worst pain possible. The outcome measure "Pain intensity" assessed as a change between baseline and post tDCS stimulation (after stimulation day 5). The calculated change in the range of positive numbers indicates decreased pain intensity post-treatment (eg. baseline 6; post treatment 4; change +2 indicating decrease of pain intensity by 2 points). Similarly, change in range of negative numbers indicates a worsening of pain intensity (eg. baseline 6; post treatment 8; change -2).
Time Frame: Assessed at baseline and post tDCS stimulation day 5
Measure: Mean (Standard Error); unit: Points on numerical rating scale
Arm/Group | Real tDCS Stimulation | Sham tDCS
Number analyzed (Participants) | 16 | 8
Points on numerical rating scale | 1.66 (0.49) | 1.60 (0.74)

ADVERSE EVENTS:
Arm/Group | Real tDCS Stimulation | Sham tDCS
Serious Adverse Events (participants affected / at risk) | 1/16 | 1/8
Other Adverse Events (participants affected / at risk) | 10/16 | 5/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Real tDCS Stimulation (N=16) | Sham tDCS (N=8)
Exacerbation of shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (2) — Exacerbation of shortness of breath and chest pain on 2 occasions in the follow-up period. Symptoms were attributed to opioid medication regimen and patient's anxiety, and the issue was resolved.
Exacerbation of Pain due to rectal cellulitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Transient change in mental status (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Real tDCS Stimulation (N=16) | Sham tDCS (N=8)
Headache (General disorders) | 2 (2) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0)
Transient Pain (General disorders) | 1 (1) | 0 (0)
Interrupted Sleep (General disorders) | 0 (0) | 1 (1)
Hypotension (General disorders) | 1 (1) | 0 (0)
Dizziness (General disorders) | 1 (1) | 0 (0)
Dry Mouth (General disorders) | 1 (1) | 0 (0)
Numbness (General disorders) | 0 (0) | 1 (1)
Worsening of Pain (General disorders) | 0 (0) | 1 (1)
Tongue tingling (General disorders) | 1 (1) | 0 (0) — Subject with diagnosis of cancer of the base of tongue; tongue tingling developed as a part of cancer treatment prior to study participation
Cellulitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Memory lapse (Nervous system disorders) | 1 (1) | 0 (0) — transient increase of memory lapse in elderly subject with history of CVA affecting frontal lobe.
Clear discharge from ear (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Urinary tract infection (Renal and urinary disorders) | 1 (1) | 0 (0)
Flu-like symptoms (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Tibial fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — tibial fracture due to mechanical fall

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes